CLINICAL TRIAL: NCT00419107
Title: Beta Cell Function in Women With Turner Syndrome
Status: Terminated | Type: Observational
Why Stopped: Completed
Sponsor: University of Aarhus (Other)
Responsible Party: Jens Sandahl Christiansen, Aarhus University Hospital, Aarhus, Denmark
Other Study IDs: 20040108
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.

SUMMARY:
Diabetes is more frequent in women with Turner syndrome. The purpose of this study is to see, in what ways the glucose metabolism is different in this study population. The hypothesis is that women with Turner Syndrome have an impaired insulin production (beta cell function).

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome

Exclusion Criteria:

* Diagnosed diabetes
* BMI>30
* Untreated cardiac or thyroid disease
* Cancer illness

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 13 women with TS and 12 control women
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2004-11; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sandahl Christiansen, prof. dr.med, Principal Investigator
Locations (1):
- Medical Department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Derived] Hjerrild BE, Holst JJ, Juhl CB, Christiansen JS, Schmitz O, Gravholt CH. Delayed beta-cell response and glucose intolerance in young women with Turner syndrome. BMC Endocr Disord. 2011 Mar 15;11:6. doi: 10.1186/1472-6823-11-6. PMID 21406078